CLINICAL TRIAL: NCT07190443
Title: Randomized Phase III Trial for Evaluating the Efficacy of Adjuvant Abemaciclib in Patients With Locoregional Recurrence of Hormone Receptor-positive, HER2-negative Breast Cancer. JCOG2313, AURA Trial.
Brief Title: Adjuvant Abemaciclib for Locoregional Recurrence of HR-positive, HER2-negative Breast Cancer (JCOG2313, AURA)
Acronym: AURA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Japanese Foundation for Cancer Research (Other)
Collaborators: Japan Clinical Oncology Group (Other)
Responsible Party: Principal Investigator, Yukinori Ozaki, Head Physician, Japanese Foundation for Cancer Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG2313; jRCTs031240666 (Other: National Cancer Center Hospital)
Record Dates: First submitted 2025-09-22; First posted 2025-09-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Locoregional Recurrence; Abemaciclib; Endocrine Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Anastrozole; exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard endocrine therapy (Arm A) (Active Comparator): Participants in Arm A will receive standard endocrine therapy alone as adjuvant treatment following curative-intent local therapy for first locoregional recurrence (LRR) of hormone receptor (HR)-positive, HER2-negative breast cancer. No CDK4/6 inhibitor is administered in this arm.
  Interventions: Drug: Endocrine Therapy (ET): letrozole, anastrozole, exemestane, tamoxifen
- Endocrine therapy in combination with abemaciclib (Arm B) (Experimental): Participants in Arm B will receive endocrine therapy in combination with abemaciclib following curative-intent local treatment for first LRR of HR-positive, HER2-negative breast cancer.
  Interventions: Drug: Endocrine therapy + Abemaciclib

INTERVENTIONS:
Drug: Endocrine therapy + Abemaciclib — This intervention consists of adjuvant endocrine therapy in combination with abemaciclib, a CDK4/6 inhibitor, administered to patients with HR-positive, HER2-negative breast cancer who have undergone curative-intent local treatment for their first LRR, including ipsilateral breast tumor recurrence, chest wall recurrence, or regional lymph node recurrence.
  Abemaciclib is given orally at a dose of 150 mg twice daily for a maximum of 2 years, in accordance with the approved dosing regimen in the adjuvant setting. The choice of endocrine therapy-aromatase inhibitor, tamoxifen, or tamoxifen plus ovarian function suppression-is determined based on menopausal status and prior treatment history.
  Arms: Endocrine therapy in combination with abemaciclib (Arm B)
Drug: Endocrine Therapy (ET): letrozole, anastrozole, exemestane, tamoxifen — This intervention consists of adjuvant endocrine therapy alone in patients with HR-positive, HER2-negative breast cancer who have undergone curative treatment for their first LRR, including ipsilateral breast tumor recurrence, chest wall recurrence, or regional lymph node recurrence.
  The choice of endocrine therapy (aromatase inhibitor, tamoxifen, or tamoxifen plus ovarian function suppression) is determined based on the patient's menopausal status and prior treatment history, as specified in the protocol. Treatment is continued for five years or until disease recurrence, unacceptable toxicity, or withdrawal of consent.
  This intervention does not include CDK4/6 inhibitors.
  Arms: Standard endocrine therapy (Arm A)

SUMMARY:
The JCOG2313 trial is a multicenter, randomized, phase III study designed to evaluate the efficacy and safety of adjuvant abemaciclib in combination with endocrine therapy versus endocrine therapy alone in patients with hormone receptor (HR)-positive, HER2-negative breast cancer who have undergone curative treatment for their first locoregional recurrence (LRR).

Although HR-positive, HER2-negative breast cancer generally has a favorable prognosis, LRR-such as ipsilateral breast tumor recurrence (IBTR), chest wall recurrence, or regional lymph node recurrence-remains a clinically significant event that increases the risk of distant metastasis. While endocrine therapy is standard in this setting, the benefit of adding chemotherapy or other agents remains unclear, and treatment strategies vary widely.

Abemaciclib, a CDK4/6 inhibitor, has shown survival benefit in the adjuvant setting for high-risk early breast cancer. However, its role in post-LRR adjuvant treatment has not been evaluated in a randomized setting. This study aims to determine whether the addition of abemaciclib to endocrine therapy can improve invasive disease-free survival (IDFS) in patients after LRR.

Eligible patients are randomized 1:1 to receive either endocrine therapy alone or endocrine therapy plus abemaciclib (150 mg twice daily for 2 years). The primary endpoint is IDFS. Secondary endpoints include distant recurrence-free survival, breast cancer-specific survival, overall survival, and safety. A total of 290 patients will be enrolled. Randomization is stratified by site of recurrence, endocrine resistance, perioperative chemotherapy, and institution.

Additionally, a prospective ancillary study will assess circulating tumor DNA (ctDNA) as a biomarker for molecular residual disease (MRD). Plasma samples will be collected at predefined time points to evaluate the prognostic and predictive value of ctDNA for relapse and treatment response.

The JCOG2313 trial addresses an unmet need in the management of HR-positive, HER2-negative LRR and may contribute to the establishment of a new standard systemic therapy and personalized monitoring strategies.

ELIGIBILITY:
Inclusion criteria:

1. The patient has been diagnosed with the first locoregional recurrence (LRR) after receiving definitive treatment for primary breast cancer. LRR includes one or more of the following:

   (i) Ipsilateral breast tumor recurrence (ii) Ipsilateral chest wall recurrence (iii) Regional lymph node recurrence
2. At least one LRR lesion must be confirmed by a biopsy, surgical specimen, or cell block from cytology, and must meet all of the following:

   (i) Pathologically confirmed as invasive breast cancer, or diagnosed as breast cancer in a cytology cell block (in cases where only a cell block is available, the initial primary breast cancer must have been invasive).

   (ii) Hormone receptor (HR) expression is positive. (iii) HER2 expression is negative.

   ※ If multiple lesions are pathologically evaluated and any lesion is HR-negative or HER2-positive, the patient is ineligible.
3. No prior diagnosis of distant metastasis of breast cancer.
4. Imaging assessment before registration confirms:

   No lymph nodes ≥10 mm in short axis No evidence of distant metastasis
5. Age ≥18 years at the time of registration.
6. ECOG Performance Status of 0 or 1.
7. Chemotherapy for LRR is allowed prior to enrollment.
8. The patient does not have bilateral breast cancer.
9. No prior history of treatment with CDK4/6 inhibitors.
10. Written informed consent has been obtained for participation in this clinical trial.

Exclusion Criteria:

1. Presence of active double cancer (synchronous malignancy requiring treatment).
2. Ongoing infectious disease requiring systemic therapy.
3. Fever ≥38.0°C at the time of registration.
4. Women who are pregnant, possibly pregnant, within 28 days postpartum, or breastfeeding; men whose partners intend to become pregnant.
5. Psychiatric illness or symptoms that interfere with daily living and may compromise trial participation.
6. Ongoing systemic administration (oral or IV) of steroids equivalent to ≥10 mg/day of prednisolone or other immunosuppressive agents.
7. Unstable angina (developed or worsened within the past 3 weeks) or myocardial infarction within the past 6 months.
8. Uncontrolled hypertension.
9. Uncontrolled diabetes mellitus despite continuous insulin or oral antidiabetic therapy.
10. Positive for HBs antigen or HCV antibodies (Patients positive for HCV antibodies are not excluded if HCV-RNA is undetectable.)
11. Positive for HIV antibodies (HIV testing is not mandatory.)
12. Presence of interstitial pneumonia, pulmonary fibrosis, or severe emphysema as diagnosed by chest CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2034-02-06 (Estimated); Study Completion 2035-02-06 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival | Up to 9 years (4 years of accrual and 5 years of follow-up)
  Defined as the time from randomization to the first occurrence of one of the following events:
  * Recurrence of invasive breast cancer in the ipsilateral breast, chest wall, or regional lymph nodes (locoregional recurrence);
  * Distant recurrence of breast cancer (metastatic disease);
  * Invasive contralateral breast cancer;
  * Second primary invasive non-breast cancer (excluding non-melanoma skin cancer and in situ cervical cancer);
  * Death from any cause. Patients who have not experienced any of the above events will be censored at the date of last disease assessment.

SECONDARY OUTCOMES:
Distant recurrence-free survival | Up to 9 years (4 years of accrual and 5 years of follow-up)
  Distant Recurrence-Free Survival (DRFS) is defined as the time from randomization to the first occurrence of distant recurrence of breast cancer or death from any cause, whichever occurs first.
  Distant recurrence is defined as radiographically or pathologically confirmed metastatic disease outside of the locoregional area.
  Patients without events will be censored at the date of last disease assessment.
  DRFS is evaluated as a secondary endpoint to assess the effectiveness of treatment in preventing distant metastatic progression.
Breast cancer-specific survival | Up to 9 years (4 years of accrual and 5 years of follow-up)
  Breast Cancer-Specific Survival (BCSS) is defined as the time from randomization to death due to breast cancer.
  Deaths from other causes (non-breast cancer-related) will be considered competing events and will be censored at the time of death.
  Patients who are alive at the time of analysis or lost to follow-up will be censored at the date of last known contact.
  BCSS is included as a secondary endpoint to evaluate the disease-specific mortality benefit of the intervention.
Overall survival | Up to 9 years (4 years of accrual and 5 years of follow-up)
  Overall Survival (OS) is defined as the time from randomization to death from any cause.
  Patients who are alive at the time of analysis or lost to follow-up will be censored at the date of last known contact.
  OS will be assessed as a secondary endpoint to evaluate the overall survival benefit of adjuvant abemaciclib in combination with endocrine therapy in the post-recurrence setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute Hospital of JFCR, Koto-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided
Plans for sharing IPD have not been finalized. Data sharing may be considered in the future pending appropriate ethical and regulatory approvals.